CLINICAL TRIAL: NCT06168201
Title: VIrtual STudy in Achondroplasia for the US (VISTA)
Acronym: VISTA
Status: Recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Collaborators: PicnicHealth (Unknown)
Responsible Party: Sponsor
Other Study IDs: 111-605
Record Dates: First submitted 2023-11-02; First posted 2023-12-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (2):
- Primary Pediatric Cohort: ≤13 years old at time of enrollment. This is an observational study.
- Secondary Adolescent and Adult Cohort: ≥14 years old at time of enrollment. This is an observational study.

SUMMARY:
This is an observational study of individuals with achondroplasia in the United States. The primary study population consists of pediatric individuals treated and untreated with VOXZOGO™. Study enrollment started in February 2023. The projected total duration of the study is approximately 5 years at minimum from start of study recruitment in February 2023, with the duration of individual prospective follow-up differing depending on the time of enrollment. The study duration may be extended based on decisions by the study sponsor.

Data will be collected in two formats for the primary pediatric study population:

1. Participant-mediated access to electronic health records(including medical imaging, when available) which will enable retrospective and prospective collection of secondary data reflecting real-life treatment use and clinical care. .
2. Primary data collection of Clinical Outcome Assessments (COAs) and questionnaire data.

Data will be collected in the following format for the adult cohort:

- Participant-mediated access to electronic health records (including medical imaging, when available) which will enable retrospective and prospective collection of secondary data reflecting real-life treatment use and clinical care.

The primary study population will include approximately 150 pediatric individuals with achondroplasia regardless of their treatment status with VOXZOGO™. Individuals may change status from untreated to treated during the prospective period of the study (or vice versa) however they will only be counted once, based on their treated status at the point of enrollment.

The secondary study population will include 20 adolescent and adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of achondroplasia
* Age at time of enrollment:

Primary Pediatric Cohort: ≤13 years old Secondary Adolescent and Adult Cohort: ≥14 years old

* Receiving medical care in the United States
* Complete PicnicHealth's onboarding process, including signing informed consent and authorization for medical record retrieval

Exclusion Criteria:

* Lack of any medical records

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The primary study population will include individuals with achondroplasia regardless of their treatment status with VOXZOGO™. Whilst individuals may change status from untreated to treated during the prospective period of the study (or vice versa), for the purposes of recruitment targets they will only be counted once, based on their treated status at the point of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Height | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
  sitting and standing measured in centimetres
Weight | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
  measured in kilograms
Body Mass Index | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
  measured in kg/m2
Head Circumference | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
  measured in centimeters
Annualized growth velocity (AGV) | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
  measured in centimeters/year
Medical diagnoses by age | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
  Clinical examination and/or radiological assessment
Surgical procedures and/or medical interventions by age | Retrospective data and prospective data for up to 5 years starting from time of study enrolment
Changes in physical functioning | every 6 months starting from time of study enrolment up to 5 years
  assessed using the Mobility and Upper Extremity Patient-Reported Outcomes Measurement Information System (PROMIS) tools
Changes in health-related quality of life (HRQoL) | every 6 months starting from time of study enrolment up to 5 years
  assessed using the Pediatric Quality of Life Inventory (PedsQL)
Adherence to treatment with VOXZOGO™ (vosoritide), if prescribed | every 6 months starting from time of study enrolment up to 5 years
  assessed using a medication adherence questionnaire to capture the number of missed doses in the prior month. Parent(ObsRO) version for all participants enrolled ages 5-13 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (7):
- United States (7):
  - UCSF, Oakland, California
  - PicnicHealth, San Francisco, California
  - Piedmont Health, Statesville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Sanford Health, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin